CLINICAL TRIAL: NCT05170529
Title: Prevalence of Non-Carious Cervical Lesions in Patient With Gingival Recession and Associated Risk Factors: A Hospital Based Cross-Sectional Study in a Sample of Adult Egyptian Dental Patients.
Brief Title: Prevalence of Non-Carious Cervical Lesions in Patient With Gingival Recession and Associated Risk Factors
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Essam Ali, Principle investigator, Cairo University
Other Study IDs: 111021
Record Dates: First submitted 2021-12-07; First posted 2021-12-28 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Non-carious Cervical Lesion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims at determining the prevalence of non carious cervical lesions in patients with gingival recession in Egyptian population and associated risk factors including gingival biotype, keratinized tissue width, gingival index, plaque index, occlusal wear grade, sensitivity. and a questionnaire will be filled by patients with another risk factors including age, gender, toothbrush frequency and type, bruxism, gastric reflux, soft drinks, alcohol and citrus fruits. Also OHIP-14 will be answered in a questionnaire form by patients.

DETAILED DESCRIPTION:
Dental patients will be recruited in a consecutive manner from diagnostic centre at Cairo University Dentistry faculty. Patients with NCCL will be selected for questionnaires and clinical examination. Thorough oral examination will be done, the full aim of the study will be explained to the patient, and patient acceptance is a must. The questionnaire will be done with face to face interview with the patient will include associated risk factors including gingival biotype, keratinized tissue width, gingival index, plaque index, occlusal wear grade, sensitivity. and a questionnaire will be filled by patients with another risk factors including age, gender, toothbrush frequency and type, bruxism, gastric reflux, soft drinks, alcohol and citrus fruits. Also OHIP-14 will be answered in a questionnaire form by patients including: functional limitations, physical pain, psychological discomfort, physical disability, psychological disability, social disability, handicap. then clinical examination will be done for NCCL using mirror, probe, light of the unit, air tip.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with NCCL and gingival recession whose age is above 15 years old
* patients consulting in dental Diagnostic Centre, faculty of dentistry, Cairo University
* patients provide informed consent

Exclusion Criteria:

* patients having problem in mouth opening or undergoing intermaxillary fixation where oral examination is not possible
* patients diagnosed with psychiatric problems

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: adult Egyptian patients with gingival recession attending the dental diagnostic centre in Cairo university
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
number of patients with non-carious cervical lesions in Egyptian adult patients with gingival recession | Day 1
  clinical examination

SECONDARY OUTCOMES:
Oral health related-quality of life (OHR-QoL) OHIP-14 questionnaire | Day 1
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt